CLINICAL TRIAL: NCT06784167
Title: Vaccine Responses in Patient With Multiple Myeloma and Non-Hodgkins Lymphoma Post CAR-T Treatment
Brief Title: Vaccine Responses in Patient With Multiple Myeloma and Non-Hodgkin Lymphoma After CAR-T Treatment
Status: Recruiting | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Amrita Desai, M.D., Principal Investigator, OHSU Knight Cancer Institute
Other Study IDs: STUDY00027998; NCI-2024-10661 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00027998 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Chronic Lymphocytic Leukemia; Diffuse Large B-Cell Lymphoma; Follicular Lymphoma; Mantle Cell Lymphoma; Multiple Myeloma; Primary Mediastinal Large B-Cell Lymphoma; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients may receive up to 3 doses of pneumococcal and/or tetanus vaccine per institutional policy of revaccination. Patients undergo blood sample collection and have medical records reviewed throughout the study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates immune responses after CAR-T therapy to find out if CAR-T therapy reduces the effectiveness of the vaccines (vaccine immunity) against diseases such as measles, mumps and rubella, among others in patients with multiple myeloma and non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess positive VPD antibody (Ab) titers prior to and at 6 months after CAR-T therapy to evaluate the impact of CAR-T on immune responses in patients undergoing CAR-T therapy.

II. To assess the change in Ab titer to S. pneumoniae and tetanus at 6 months and 1 year post-vaccination and evaluate if titer increases are correlated to post-vaccination CD4+ count and IgG level.

OUTLINE: This is an observational study.

Patients may receive up to 3 doses of pneumococcal and/or tetanus vaccine per institutional policy of revaccination. Patients undergo blood sample collection and have medical records reviewed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* * Willingness to provide written informed consent before any study-specific procedures or activities are performed

  * Age ≥ 18 years of age, at the time of consent
  * Documented, histologically or cytologically confirmed diagnosis of multiple myeloma (MM), diffuse large B cell lymphoma (DLBCL),follicular lymphoma (FL), mantle cell lymphoma (MCL), chronic lymphocytic leukemia (CLL), or small lymphocytic lymphoma (SLL), or primary mediastinal B cell lymphoma (PMBL). All number of prior lines of therapy are allowed
  * History of prior vaccination against common VPD
  * Approved by managing physician for CAR-T therapy, with preparative conditioning planned within the next 90 days
  * Approved by managing physician for revaccination against Streptococcus pneumoniae or tetanus

Exclusion Criteria:

* * Ongoing use of immunosuppressive agents or plans for immunosuppressive therapy that would interfere with interpretation of study endpoints

  * Uncontrolled, intercurrent illness including, but not limited to, systemic infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements or make the study procedures unadvisable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple myeloma and non-hodgkin lymphoma recruited through OHSU Knight Cancer Institute
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-01-11 (Estimated); Study Completion 2027-04-12 (Estimated)

PRIMARY OUTCOMES:
Preserved immunity | Up to 12 months after CAR-T cell infusion
  Will be defined as titers that meet the definition of positive both pre- and post-CAR-T cell infusion. The proportion of subjects who have preserved immunity to each VPD will be estimated with an exact 95% confidence interval.

SECONDARY OUTCOMES:
Change in antibody titers | At baseline, at 6 months and at 1 year after vaccination
  Immune reconstitution will be reported based on ELISA assays for S. pneumoniae or tetanus after each dose of respective vaccine for the re-vaccination populations. Will be correlated with the changes of CD4+ and IgG using a Spearman correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Desai, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States